CLINICAL TRIAL: NCT06436742
Title: A Phase 1b, Double-Blinded, Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Efficacy of ARGX-119 in Adult Participants With DOK7-Congenital Myasthenic Syndromes
Brief Title: A Phase 1b Study to Investigate Safety and Tolerability of ARGX-119 in Adult Participants With DOK7-Congenital Myasthenic Syndromes (CMS)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-119-2302; 2023-509872-41-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-21; First posted 2024-05-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Congenital Myasthenic Syndrome; CMS
MeSH Terms: conditions — Myasthenic Syndromes, Congenital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-blinded treatment period - ARGX-119 IV (Experimental): Participants receive ARGX-119 during the double-blinded treatment period
  Interventions: Biological: ARGX-119
- Double-blinded treatment period - Placebo IV (Placebo Comparator): Participants receive placebo during the double-blinded treatment period
  Interventions: Other: Placebo
- Active-treatment period - ARGX-119 IV (Experimental): Participants receive ARGX-119 during the active-treatment period
  Interventions: Biological: ARGX-119

INTERVENTIONS:
Biological: ARGX-119 — Intravenous infusion of ARGX-119
  Arms: Active-treatment period - ARGX-119 IV; Double-blinded treatment period - ARGX-119 IV
Other: Placebo — Intravenous infusion of placebo
  Arms: Double-blinded treatment period - Placebo IV

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ARGX-119 in adult participants with DOK7- Congenital Myasthenic Syndromes. The study will also assess how ARGX-119 is processed by the body (pharmacokinetics), how the immune system reacts to it (immunogenicity), and how it may improve the way patients feel and function.

After the screening period, eligible participants will be randomized in a 4:1 ratio to receive intravenous infusions of ARGX-119 or placebo during the double-blinded treatment period. Participants will then enter the follow-up period. After the follow-up period, participants may enrol in the active-treatment period, where they will receive open-label ARGX-119.

The full duration of the study is approximately 38 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Has genetically confirmed congenital myasthenic syndromes due to mutation of downstream of kinase 7 (DOK7-CMS).
* Participants taking oral beta agonists (eg, albuterol, salbutamol, ephedrine) must have been receiving the medication for more than 3 months and agree to remain on a same stable dosing regimen of the same medication until the end of the study.

Exclusion Criteria:

* Diagnosis of CMS due to mutation of any gene other than DOK7.
* Known medical condition that would interfere with an accurate assessment of CMS, confound the results of the study, or put the patient at undue risk, as assessed by the investigator.
* History of malignancy, cancer, unless considered cured by adequate treatment with no evidence of recurrence for more than 5 years. Adequately treated participants with the following cancers can be included at any time: Basal cell or squamous cell skin cancer, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histological findings of prostate cancer.
* Pregnant or lactating state or intention to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-08-24 (Estimated); Study Completion 2028-01-24 (Estimated)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs) | Up to week 42
Change from active-treatment baseline over time for 6MWT distance | Up to 72 weeks
  The 6-minute walk test (6MWT) measures the distance a participant walks in 6 minutes. Before and after the 6MWT assessment, the participant's blood pressure, heart rate, and SPO2 will be recorded, and the participant's perception of fatigue and dyspnea will be measured.

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of ARGX-119 | Up to 42 weeks + 72 weeks
Incidence of ADA against ARGX-119 | Up to 42 weeks + 72 weeks
  ADA : anti-drug antibodies
Change from baseline over time for key components of the QMG scale | Up to 42 weeks + 72 weeks
  The Quantitative Myasthenia Gravis (QMG) scale is a standardized quantitative scoring system that was developed to assess disease severity based on impairment of body function and structures in patients with MG. Minimum value: 0 (no disease severity); Maximum value: 39 (highest disease severity). The change from active-treatment baseline will be used for the 72 week timepoint.
Change from baseline over time for MG-ADL | Up to 42 weeks + 72 weeks
  The Myasthenia Gravis Activities of Daily Living (MG-ADL) is an 8-item scale that assesses MG symptoms and their effects on daily activities. Minimum value: 0 (normal symptoms); Maximum value: 24 (most severe symptoms). The change from active-treatment baseline will be used for the 72 week timepoint.
Change from baseline over time for PROMIS-GH scale | Up to 42 weeks
  The Patient-Reported Outcomes Measurement Information System Global Health (PROMIS-GH) is a 10-item participant completed quality of life questionnaire that measures global physical health and mental health. The participant records their response to each question on a 5-point Likert scale, with lower scores indicating poorer health (Minimum value: 0, Maximum value: 20)
Change from active-treatment baseline over time for 6MWT cadence | Up to 72 weeks
  The 6-minute walk test (6MWT) measures the distance a participant walks in 6 minutes. Before and after the 6MWT assessment, the participant's blood pressure, heart rate, and SPO2 will be recorded, and the participant's perception of fatigue and dyspnea will be measured.
Change from active-treatment baseline over time for PROMIS PF-WMA-SF | Up to 72 weeks
  The PROMIS PF-WMA-SF is an 11-item, participant-completed questionnaire that assesses lower and upper extremity function and associated activities of daily living. The questionnaire asks the participant to rate the items on a 5-point scale of 5 (without any difficulty) to 0 (unable to do).
Change from active-treatment baseline over time for Neuro-QoL fatigue | Up to 72 weeks
Change from active-treatment baseline over time for FVC | Up to 72 weeks
Change from active-treatment baseline over time for PGI-C | Up to 72 weeks
Change from active-treatment baseline over time for PGI-S | Up to 72 weeks
Change from active-treatment baseline over time for CGI-C | Up to 72 weeks
Change from active-treatment baseline over time for CGI-S | Up to 72 weeks
Change from active-treatment baseline over time for EQ-5D-5L | Up to 72 weeks
Incidence of AEs and SAEs | Up to 72 weeks
  AE : Adverse events ; SAE : Serious Adverse events

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - UC Davis Medical Center, Sacramento, California
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
- Ottawa Hospital Research Institute - Civic Campus, Ottawa, Canada
- France (2):
  - CHU - Hospital de la Timone, Marseille
  - Group Hospitalier Pitie-Salpetriere, Paris
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy
- Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia, Spain
- United Kingdom (2):
  - Clinical Trials Centre - South Eastern Health and Social Care Trust - The Ulster Hospital, Belfast
  - John Radcliffe Hospital - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No